CLINICAL TRIAL: NCT06702527
Title: Optimizing Clinical Outcomes in Patients Undergoing M-TEER for Severe Functional Mitral Regurgitation Towards Improved Guideline-directed Medical Therapy - The MOTOR Registry
Brief Title: Optimizing Clinical Outcomes in Patients Undergoing Mitral Transcatheter Edge-to-edge Repair (M-TEER) for Severe Functional Mitral Regurgitation Towards Improved Guideline-directed Medical Therapy
Acronym: MOTOR
Status: Not yet recruiting | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Responsible Party: Sponsor
Other Study IDs: The MOTOR Registry
Record Dates: First submitted 2024-11-19; First posted 2024-11-25 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Mitral Regurgitation Functional; Heart Failure; M-TEER
Keywords: Mitral Regurgitation; Heart Failure; M-TEER; Optimizing GDMT; Functional Mitral Regurgitation
MeSH Terms: conditions — Heart Failure; Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- M-TEER patients: Patients with optimized guideline-directed medical therapy (GDMT) undergoing mitral transcatheter edge-to-edge repair (M-TEER, using the PASCAL system) for severe functional mitral regurgitation.
  Interventions: Procedure: Mitral transcatheter edge-to-edge repair

INTERVENTIONS:
Procedure: Mitral transcatheter edge-to-edge repair — Mitral transcatheter edge-to-edge repair with the PASCAL system
  Other Names: M-TEER

SUMMARY:
A multi-centre, prospective, observational pilot registry in patients undergoing mitral valve repair for severe functional mitral regurgitation to report the heart failure drug therapy and dosing before the mitral valve procedure and afterwards to assess whether the recommended maximal dose of medication is administered. This maximal dose, although recommended, might not be tolerated well by patients and can cause side-effects. Researchers will determine whether the mitral valve repair procedure might have a possible effect on increasing the drug therapy towards the recommended optimal doses.

DETAILED DESCRIPTION:
Mitral transcatheter edge-to-edge repair (M-TEER) has become an important therapy in the management of severe functional mitral regurgitation (FMR).

These patients often have left ventricular dilatation with associated left ventricular failure and undergo intervention after guideline-directed medical therapy (GDMT) is optimised.

However, many patients cannot tolerate maximal doses of these drugs, some of which are potent vasodilators, due to the potential for hypotension and other side effects.

After M-TEER, with significant reduction of valve regurgitation, and a consequent improvement in systemic blood pressure and left ventricular function, it may be possible to further optimize GDMT and thus improve patients' clinical outcomes.

This pilot registry will be conducted in up to 4 German centres with a minimum annual volume of ~ 50 M-TEER procedures aiming for an environment of 100 patients.

This registry aims to:

* document the extent of suboptimal GDMT in patients undergoing M-TEER for severe FMR and to assess the potential to improve care towards maximal recommended medical therapy.
* compare 6- and 12-months heart failure (HF) hospitalization post-procedure compared to 12- and 6-months historical HF hospitalisation prior the index procedure. Functional status (NYHA class, 6-minute walk test) to be assessed at baseline and at 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* mitral transcatheter edge-to-edge repair (M-TEER) patients treated with the PASCAL system (≥ 18 years) as per the current approved indication and local Heart Team decision
* Severe functional and mixed-type mitral regurgitation with LV-EF < 50%
* Patient with optimized guideline-directed medical therapy (GDMT): A minimum of 3 points in the pre-defined GMDT scoring system
* Provision of written informed consent

Exclusion Criteria:

* Degenerative mitral regurgitation
* Emergency procedure
* Re-do or concomitant (mitral/tricuspid) procedures
* Patients on maximum dose GDMT
* Atrial functional mitral regurgitation (FMR)
* Coronary revascularisation within the last 3 months
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe functional and mixed-type mitral regurgitation with optimized GMDT undergoing M-TEER (using the PASCAL system)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Heart Failure hospitalizations after mitral transcatheter edge-to-edge repair (M-TEER) | 6 and 12 months
  Number of 6- and 12-months heart failure (HF) hospitalizations post M-TEER procedure compared to 12- and 6-months historical HF hospitalization prior the index procedure

SECONDARY OUTCOMES:
New York Heart Association (NYHA) class | 6 months
  NYHA class at baseline and 6-months follow-up
6-minute walk test | 6 months
  6-minute walk test at baseline and 6-months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Malte Sinning, Prof., Principal Investigator — Cellitinnen Hospital St. Vinzenz
Locations (1):
- Cellitinnen Hospital St. Vinzenz, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
no IPD shared with other researchers, sponsor owns database

REFERENCES:
- [Background] Stone GW, Abraham WT, Lindenfeld J, Kar S, Grayburn PA, Lim DS, Mishell JM, Whisenant B, Rinaldi M, Kapadia SR, Rajagopal V, Sarembock IJ, Brieke A, Marx SO, Cohen DJ, Asch FM, Mack MJ; COAPT Investigators. Five-Year Follow-up after Transcatheter Repair of Secondary Mitral Regurgitation. N Engl J Med. 2023 Jun 1;388(22):2037-2048. doi: 10.1056/NEJMoa2300213. Epub 2023 Mar 5. PMID 36876756
- [Background] Greene SJ, Butler J, Albert NM, DeVore AD, Sharma PP, Duffy CI, Hill CL, McCague K, Mi X, Patterson JH, Spertus JA, Thomas L, Williams FB, Hernandez AF, Fonarow GC. Medical Therapy for Heart Failure With Reduced Ejection Fraction: The CHAMP-HF Registry. J Am Coll Cardiol. 2018 Jul 24;72(4):351-366. doi: 10.1016/j.jacc.2018.04.070. PMID 30025570
- [Background] Savarese G, Bodegard J, Norhammar A, Sartipy P, Thuresson M, Cowie MR, Fonarow GC, Vaduganathan M, Coats AJS. Heart failure drug titration, discontinuation, mortality and heart failure hospitalization risk: a multinational observational study (US, UK and Sweden). Eur J Heart Fail. 2021 Sep;23(9):1499-1511. doi: 10.1002/ejhf.2271. Epub 2021 Jun 28. PMID 34132001
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Adamo M, Tomasoni D, Stolz L, Stocker TJ, Pancaldi E, Koell B, Karam N, Besler C, Giannini C, Sampaio F, Praz F, Ruf T, Pechmajou L, Neuss M, Iliadis C, Baldus S, Butter C, Kalbacher D, Lurz P, Melica B, Petronio AS, von Bardeleben RS, Windecker S, Butler J, Fonarow GC, Hausleiter J, Metra M. Impact of Transcatheter Edge-to-Edge Mitral Valve Repair on Guideline-Directed Medical Therapy Uptitration. JACC Cardiovasc Interv. 2023 Apr 24;16(8):896-905. doi: 10.1016/j.jcin.2023.01.362. Epub 2023 Mar 22. PMID 37100553